CLINICAL TRIAL: NCT04402957
Title: Multicenter, Randomized, Double-Blind, Placebo-Controlled, Proof of Concept Study of LSALT Peptide as Prevention of Acute Respiratory Distress Syndrome (ARDS) and Acute Kidney Injury in Patients Infected With SARS-CoV-2 (COVID-19)
Brief Title: LSALT Peptide vs. Placebo to Prevent ARDS and Acute Kidney Injury in Patients Infected With SARS-CoV-2 (COVID-19)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arch Biopartners Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AB002
Record Dates: First submitted 2020-05-12; First posted 2020-05-27 (Actual); Results first posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: COVID; Severe Acute Respiratory Syndrome; Sars-CoV2; Acute Kidney Injury; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; Acute Kidney Injury; Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 100 mL drug-free IV saline infusion over 2 hours daily
  Interventions: Drug: Placebo
- LSALT (Experimental): 100 mL of 5 mg IV LSALT peptide infusion over 2 hours daily
  Interventions: Drug: LSALT peptide

INTERVENTIONS:
Drug: LSALT peptide — LSALT, a peptide drug with the sequence NH3-LSALTPSPSWLKYKAL-COOH, binds to dipeptidase-1 (DPEP-1) but does not inhibit its biologic enzymatic activity. LSALT peptide inhibits leukocyte recruitment in multiple experimental disease models through the direct inhibition of leukocyte adhesion to DPEP-1 present in lungs, kidney, and liver.
  Other Names: Metablok
  Arms: LSALT
Drug: Placebo — 0.9% saline solution
  Arms: Placebo

SUMMARY:
To evaluate the proportion of subjects alive and free of respiratory failure (e.g. need for non-invasive or invasive mechanical ventilation, high flow oxygen, or ECMO) and free of the need for continued renal replacement therapy (RRT) on Day 28. The need for continued RRT at Day 28 will be defined as either dialysis in the past 3 days (Day 26, 27, or 28) or an eGFR on Day 28 <10 mL/min/1.73 m2.

DETAILED DESCRIPTION:
This study is a parallel group, randomized, third-party blinded, multicenter study to assess safety and efficacy of LSALT peptide versus placebo in hospitalized patients with confirmed infection or recent confirmed infection with complications associated with COVID-19. Following screening and after establishing baseline parameters such as lung and renal function, clinical chemistries, coagulation, hematology, and urinalysis, and satisfying all inclusion and exclusion criteria, patients will be randomized to one of two blinded treatment regimens:

1. 100 mL of 5 mg IV LSALT peptide infusion over 2 hours daily
2. 100 mL drug-free IV saline infusion over 2 hours daily.

Thirty (30) patients will be randomized to active drug (LSALT peptide) and 30 patients will be randomized to matching placebo. This study will be third-party blind with only the Pharmacist at the site unblinded for the purpose of preparing drug/placebo for injection.

Patients will be followed for safety and efficacy up to Day 28, with Day 1 being the day of randomization to assess safety. After assessing the risk of ARDS and satisfying all inclusion and exclusion criteria, the patient will be randomized to 5 mg LSALT peptide or blinded placebo to be given intravenously once daily for a maximum of 14 days. Physical and respiratory examinations, vital signs, and adverse events will be recorded throughout the study, including Day 28 (EOS). Blood chemistries, hematology, coagulation, urinalysis, ECG, SARS-CoV-2 tests, eGFR, and chest x-ray (CXR) will be assessed at Day 1 (Screening/Baseline) prior to initiation of study drug, and on Day 3, EOT, and at EOS, as well as when clinically indicated. The ECG at EOS will only be obtained if clinically indicated. An additional CXR will be obtained at time of clinical improvement. Cytokines/biomarkers and pharmacokinetics (PK) will be assessed at Day 1 (Screening/Baseline) prior to initiation of study drug, at 1 (mid-dose) and 2 hours (end of infusion) of drug therapy on Days 1, 3, EOT, and a single blood sample at EOS for cytokines/biomarkers only. Where applicable, a urinary pregnancy test will be obtained at Screening in women of childbearing potential. Questionnaires (APACHE II, SOFA) will be obtained at Baseline, Day 3, EOT, and EOS; venous blood gas (VBG) or HCO3 (bicarbonate) levels may be substituted for arterial blood gas (ABG) if it is considered standard-of-care (SOC) or in the patient's best interest, and results in comparable APACHE II and SOFA scores. Other questionnaires (Berlin Definition and modified Medical Research Council Dyspnea Scale) will be assessed at Baseline, Day 3, EOT, and EOS. IgG, IgA, and IgM antiviral antibodies will be collected at Baseline and EOS. Patients will be maintained on the SOC per institutional guidelines, including prophylaxis or treatment of VTE, throughout the study.

A Data and Safety Monitoring Board (DSMB) will evaluate patients on a continuing basis for primarily safety assessments. Per the DSMB Charter, the DSMB will meet at least monthly if not more frequently based upon enrollment throughout the study period.

ELIGIBILITY:
Inclusion Criteria (Amendment 3, 15FEB2021):

1. Male and female hospitalized patients between 18 and 80 years of age at time of consent.
2. Clinical and laboratory diagnosis of COVID-19 infection. Patients must be positive for the SARS-CoV-2 by Real-Time Reverse Transcriptase (RT)-PCR

   Diagnostic Panel or have an existing complication secondary to SARS-CoV-2 infection which was positive within 2 weeks of entry into the study. Further, patients must have at least two of the following three symptoms:
   * Fever (oral temperature ≥ 100.4 °F [> 38 °C]) with or without chills
   * Dyspnea or difficulty breathing (≤ 2 on mMRC dyspnea scale)
   * Nonproductive cough
   * Or other signs and symptoms of established complications to SARS-CoV-2 infection (e.g. coagulopathy, cardiomyopathy, acute kidney injury, and/or acute liver injury) within the limits of Exclusion Criteria 8
3. Patients must present with moderate to severe illness as defined below:

   * Moderate illness: Patients who have evidence of lower respiratory disease by clinical assessment or imaging and an oxygen saturation (SpO2) > 93% on room air at sea level
   * Severe illness: Patients who have a respiratory frequency > 30 breaths per minute (bpm), SpO2 ≤ 93% on room air at sea level, ratio of arterial partial pressure of oxygen to fraction of inspired oxygen (PaO2/FiO2) < 300, or lung infiltrates > 50%.
4. APACHE II score < 20 or establishment of survivability of the patient beyond 48 hours following randomization
5. Therapies which have been shown to be beneficial and are included in standard COVID-19 treatment guidelines (e.g. those of WHO or NIH, or institutional guidelines) are permitted
6. Sexually active women of child-bearing potential (WCBP) must be using a medically acceptable method of birth control throughout the study and for at least 1 day following the end of study, and have a negative urine pregnancy test at the Screening visit. A WCBP is defined as a female who is biologically capable of becoming pregnant. A medically acceptable method of birth control includes intrauterine devices in place for at least 3 months, surgical sterilization, or the implant. In patients who are not sexually active, abstinence is an acceptable form of birth control and urine will be tested per protocol. Women who are of nonchild-bearing potential, i.e., post-menopause, must have this condition captured in their medical history. Pregnant women and nursing mothers are excluded from this study.
7. Patient or LAR is available and willing to give written informed consent, after being properly informed of the nature and risks of the study and prior to engaging in any study-related procedures.

Exclusion Criteria:

1. Known sensitivity, allergy, or previous exposure to LSALT peptide.
2. Exposure to any investigational drug or device <90 days prior to entry into study.
3. Treatment with immunomodulators or immunosuppressant drugs, including but not limited to IL-6 inhibitors, TNF inhibitors, anti-IL-1 immunomodulators, and JAK inhibitors within five half-lives or 30 days (whichever is longer) prior to randomization and throughout the study period. However, should any of these treatments become standard-of-care and incorporated into clinical treatment guidelines (e.g. those of WHO or NIH), the treatment is permitted. Further, low-dose oral prednisone (<20 mg/day) and inhaled steroids (e.g. treatment of asthma) are allowed in the study.
4. Anticipated transfer to another hospital or medical center within 72 hours, which is not a study site.
5. Uncontrolled of poorly treated active hepatitis B (HBV), hepatitis C (HepC), or HIV infection. Those subjects who are positive for HBV, HepC, or HIV but are well-controlled with low viral loads are allowed to participate in this study:

   * HBV low viral load defined as <20,000 IU/mL
   * HepC low viral load defined as <800,000 IU/mL
   * HIV low viral load defined as <5000 copies/mL
6. Participation in another drug or device study at any time during this study, for example:

   * Ulinastatin 200,000 IU or greater
   * High dose intravenous Vitamin C
   * Budesonide and formoterol
   * Bevacizumab to prevent ARDS
   * Dornase alfa to reduce hypoxemia in ventilated trauma patients.
7. As indicated in the inclusion criteria, pregnant female patients are excluded from study. Further, female patients who are nursing are excluded from study.
8. Has any medical condition considered to be clinically significant and could potentially affect patient safety or study outcome, including but not limited to:

   * Acute or chronic kidney disease (stage-4 or -5 renal impairment; eGFR<30 mL/min/1.73 m2 or hemodialysis)
   * End-stage malignancy undergoing treatment
   * Immunocompromised patients or those with medical/surgical conditions (e.g., solid organ transplantation) which require chronic immunosuppression
   * Chronic hematologic disease which, in the opinion of the PI, prohibits the patient from entering into study
   * Acute liver injury with AST and/or ALT levels greater than 3x ULN unless recent injury (within 2 weeks) likely due to COVID-19 infection
   * History of coagulopathy within the last year as defined by abnormal ACT, aPTT, and/or PT/INR values at least 2-fold outside normal limits, and currently present at screening, and/or
   * End-stage lung disease, acute lung injury, severe chronic obstructive pulmonary disease (COPD) as assessed by the GOLD criteria (GOLD Stage IV), or mechanical ventilation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2021-05-27 (Actual); Study Completion 2022-06-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (3):
  - VA San Diego Healthcare System, San Diego, California
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - LSU Health Shreveport, Shreveport, Louisiana
- Canada (2):
  - University of Calgary - Foothills Medical Centre, Calgary, Alberta
  - University of Calgary - Peter Lougheed Centre, Calgary, Alberta
- Turkey (Türkiye) (2):
  - Ankara City Hospital, Ankara
  - Istanbul University Cerrahpasa, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Somayaji R, Luke DR, Lau A, Guner R, Tabak OF, Hepokoski M, Gardetto N, Conrad SA, Kumar SD, Ghosh K, Robbins SM, Senger DL, Sun D, Lim RKS, Liu J, Eser F, Karaali R, Tremblay A, Muruve D. Multicentre, randomised, double-blind, placebo-controlled, proof of concept study of LSALT peptide as prevention of acute respiratory distress syndrome and acute kidney injury in patients infected with SARS-CoV-2 (COVID-19). BMJ Open. 2024 Mar 15;14(3):e076142. doi: 10.1136/bmjopen-2023-076142. PMID 38490660

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | LSALT
Started | 31 | 30
Completed | 29 | 29
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | LSALT | Total
Number analyzed (Participants) | 31 | 30 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (10.24) | 62.3 (8.71) | 59.8 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 20 | 21 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 5 | 7
  White | 26 | 22 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m2] | 32.29 (10.064) | 31.72 (5.571) | 32.04 (8.366)
Chronic Lung Disease [Count of Participants; unit: Participants] | 3 | 5 | 8
Chronic Renal Disease [Count of Participants; unit: Participants] | 1 | 1 | 2
Cardiovascular Disease [Count of Participants; unit: Participants] | 15 | 18 | 33
Diabetes [Count of Participants; unit: Participants] | 10 | 13 | 23
PaO2/FiO2 Ratio [Mean (Standard Deviation); unit: mmHg] | 247.956 (93.762) | 247.097 (111.3844) | 247.527 (106.728)

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Proportion of Subjects Alive and Free of Respiratory Failure and Free of the Need for Continued Renal Replacement Therapy (RRT) on Day 28 (as Per Protocol AB002 - Version 1, Dated 09JUNE2020)
Description: Respiratory failure is defined as the need for non-invasive or invasive mechanical ventilation, high flow oxygen [≥ 6 L/minute], or ECMO. The need for continued RRT at Day 28 will be defined as either dialysis in the past 3 days (Day 26, 27, or 28) or an eGFR on Day 28 <10 mL/min/1.73 m2.
Time Frame: 28 days
Population: The primary efficacy endpoint was the proportion of patients alive and free of respiratory failure (need for non-invasive or invasive mechanical ventilation, high flow oxygen, or ECMO) and free of the need for continued RRT on Day 28.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | LSALT
Number analyzed (Participants) | 31 | 30
Participants | 28 | 28

2. Secondary Outcome: All-cause Mortality
Time Frame: 28 days
Population: The all-cause mortality rate within 28 days from randomization was compared between the treatment groups using a CMH test.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | LSALT
Number analyzed (Participants) | 31 | 30
Participants | 0 | 1

3. Secondary Outcome: The Presence of and Severity of ARDS as an Ordinal Outcome of the Proportion of Patients Who Have None, Mild, Moderate, or Severe ARDS
Time Frame: 28 days
Population: Number of patients with ARDS on Day 28 (EOS).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | LSALT
Number analyzed (Participants) | 31 | 30
Participants
  Mild ARDS | 1 | 1
  Moderate ARDS | 0 | 0
  Severe ARDS | 1 | 1
  No ARDS | 29 | 28

4. Secondary Outcome: Time to Each of Mild, Moderate, or Severe ARDS
Time Frame: 28 days
Population: The proportion of patients that will develop ARDS at a given time point in the study.
Measure: Number; unit: proportion of participants
Arm/Group | Placebo | LSALT
Number analyzed (Participants) | 31 | 30
proportion of participants
  Day 3 | 0.13 | 0.1
  Day 14 | 0.2 | 0.13
  Day 28 | 0.2 | 0.13

5. Secondary Outcome: The Number of Ventilation-free Days
Time Frame: 28 days
Population: Comparison of ventilation-free days in placebo and LSALT treated patients.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | LSALT
Number analyzed (Participants) | 31 | 30
days | 20.9 (9.94) | 22.8 (7.34)

6. Secondary Outcome: Time on Nasal Cannula or Oxygen Mask
Time Frame: 28 days
Population: Only patients that were on nasal cannula or oxygen mask were analysed.
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | Placebo | LSALT
Number analyzed (Participants) | 20 | 17
hours | 203.6 [88 to 319.2] | 192.1 [43.3 to 340.9]

7. Secondary Outcome: Length of Stay in ICU and Hospital (Admission to Discharge)
Time Frame: 28 days
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | LSALT
Number analyzed (Participants) | 31 | 30
days
  Length of stay in hospital | 9 [3 to 28] | 9.5 [4 to 28]
  Length of stay in ICU | 0 [0 to 0] | 0 [0 to 0]

8. Secondary Outcome: Virologic Clearance Rate
Description: SARS-CoV2 testing by swab (nasopharyngeal, nasal, throat, sputum, or lower respiratory tract) at baseline (Day 1) and every 3 days thereafter until eradication
Time Frame: 28 days
Population: The virologic clearance rate (proportion of patients with a negative test result) at day 28 (EOS).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | LSALT
Number analyzed (Participants) | 31 | 30
Participants | 21 | 17

9. Secondary Outcome: Worst PaO2/FiO2 Ratio Following Enrollment
Description: The worst change in PaO2/FiO2 ratio from baseline (Day 1) over the course of the study was analyzed in patients. A negative value indicates a decrease in PaO2/FiO2 ratio compared to baseline.
Time Frame: 28 days
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Placebo | LSALT
Number analyzed (Participants) | 31 | 30
mmHg | -175.9 [-447.62 to 411.90] | -200.89 [-410.71 to 183.18]

10. Secondary Outcome: Change in PaO2/FiO2 Ratio
Time Frame: 28 days
Population: Change from baseline to day 28 (EOS) in PaO2/FiO2 ratio.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | LSALT
Number analyzed (Participants) | 31 | 30
mmHg | -25.708 (254.6656) | -141.217 (169.476)

11. Secondary Outcome: Change in Baseline Modified Medical Research Council (mMRC) Score
Description: Change in modified Medical Research Council score (0 to 4) with 4 being the most severe outcome. This scale is used to assess the degree of baseline functional disability due to dyspnea.
Time Frame: 28 days
Population: Change from baseline to day 28 (EOS) of modified Medical Research Council score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | LSALT
Number analyzed (Participants) | 28 | 27
score on a scale | -1 (1.12) | -1.4 (1.01)

12. Secondary Outcome: Change in Acute Physiologic Assessment and Chronic Health Evaluation (APACHE) II Score
Description: Change in APACHE II score (0 to 71) with 71 being the most severe outcome
Time Frame: 28 days
Population: Change from baseline to day 28 (EOS) in APACHE II score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | LSALT
Number analyzed (Participants) | 24 | 21
score on a scale | -0.8 (4.39) | -1.9 (3.87)

13. Secondary Outcome: Change in Daily Sequential Organ Failure Assessment (SOFA) Score From Baseline in Patients With Extrapulmonary Organ Dysfunction
Description: Change in SOFA score (0 to 4) with 4 being the most severe outcome
Time Frame: 28 days
Population: A comparison of change from baseline in SOFA score. A negative value indicates a decrease in SOFA score compared to the baseline.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Placebo | LSALT
Number analyzed (Participants) | 24 | 21
score on a scale | -1.2 [-4 to 3] | -0.7 [-4 to 3]

14. Secondary Outcome: Change in Liver Function by Alanine Aminotransferase (ALT) Test
Description: ALT measured in IU/L
Time Frame: 28 days
Population: Change from baseline liver function by ALT.
Measure: Mean (95% Confidence Interval); unit: IU/L
Arm/Group | Placebo | LSALT
Number analyzed (Participants) | 31 | 30
IU/L | -1.4 [-14.3 to 11.4] | -5.9 [-19 to 7.2]

15. Secondary Outcome: Change in Liver Function by Aspartate Transferase (AST) Test
Description: AST measured in IU/L
Time Frame: 28 days
Population: Change from baseline in liver function by AST.
Measure: Mean (95% Confidence Interval); unit: IU/L
Arm/Group | Placebo | LSALT
Number analyzed (Participants) | 31 | 30
IU/L | -19.4 [-28.9 to -9.9] | -15.4 [-25.3 to -5.5]

16. Secondary Outcome: Change in Liver Function by Total Bilirubin Test
Description: Total bilirubin measured in umol/L
Time Frame: 28 days
Population: Change from baseline in liver function by bilirubin.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Placebo | LSALT
Number analyzed (Participants) | 31 | 30
umol/L | 2.8112 (5.47094) | -1.0602 (5.52912)

17. Secondary Outcome: Change in Renal Function by Serum Creatinine (SCr) Test
Description: SCr measured in umol/L
Time Frame: 28 days
Population: Change in serum creatinine from baseline at day 28 (EOS)
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Placebo | LSALT
Number analyzed (Participants) | 28 | 28
umol/L | -1.463 (16.6250) | -1.664 (15.4972)

18. Secondary Outcome: Change in Activated Coagulation Time (ACT)
Description: ACT measured in seconds
Time Frame: 28 days
Population: Change from baseline to day 28 (EOS) in prothrombin time (PT).
Measure: Mean (Standard Deviation); unit: sec
Arm/Group | Placebo | LSALT
Number analyzed (Participants) | 21 | 16
sec | 0.0991 (2.79345) | -0.7688 (0.82439)

19. Secondary Outcome: Change in Activated Partial Thromboplastin Time (aPTT)
Description: aPTT measured in seconds
Time Frame: 28 days
Population: Change from baseline to day 28 (EOS) in aPTT.
Measure: Mean (Standard Deviation); unit: sec
Arm/Group | Placebo | LSALT
Number analyzed (Participants) | 25 | 24
sec | 2.232 (9.43189) | 1.4667 (5.21783)

20. Secondary Outcome: Change in Prothrombin International Normalized Ratio (INR)
Time Frame: 28 days
Population: Change from baseline to day 28 (EOS) in prothrombin INR.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Placebo | LSALT
Number analyzed (Participants) | 27 | 24
ratio | 0.0331 (0.29399) | -0.0658 (0.08495)

21. Secondary Outcome: Vasopressor-free Days
Time Frame: 28 days
Population: The data are not reported because testing for this specific measure was not run as the clinical sites did not have the ability/means to perform the assessment. Additionally, there are no plans to collect or analyze the data in the future.
Arm/Group | Placebo | LSALT
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Change From Maximal Radiographic Damage to EOT
Time Frame: 28 days
Population: as for outcome 21
Arm/Group | Placebo | LSALT
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Change in Renal Function by Estimated Glomerular Filtration Rate (eGFR) Test
Description: eGFR measured in ml/min/1.73m2
Time Frame: 28 days
Population: as for outcome 21
Arm/Group | Placebo | LSALT
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: Change in Hs-troponin Levels
Time Frame: 28 days
Population: as for outcome 21
Arm/Group | Placebo | LSALT
Number analyzed (Participants) | 0 | 0

25. Secondary Outcome: Change in Antiviral IgG, IgA, and IgM Levels
Description: Immunoglobulins measured in mg/dL
Time Frame: 28 days
Population: as for outcome 21
Arm/Group | Placebo | LSALT
Number analyzed (Participants) | 0 | 0

26. Other Pre Specified Outcome: Health Outcomes Endpoint: Total Healthcare Costs From Admission to Discharge Between Treatment Groups
Time Frame: 28 days
Population: Healthcare costs were not analyzed in this study.
Arm/Group | Placebo | LSALT
Number analyzed (Participants) | 0 | 0

27. Other Pre Specified Outcome: Exploratory Endpoint: Change in Serum Cytokines Including IL-1a, IL-1b, and Ferritin Levels as Well as Other Exploratory Biomarkers Drawn at the Same Time as LSALT Peptide Concentrations
Description: Fold change from baseline cytokines measured in ng/mL
Time Frame: 28 days
Population: Fold change in serum cytokine levels from baseline to day 28 (EOT).
Measure: Median (Inter-Quartile Range); unit: foldchange
Arm/Group | Placebo | LSALT
Number analyzed (Participants) | 25 | 25
foldchange
  CCL7 | 0.67 [0.3 to 1.01] | 0.62 [0.25 to 0.97]
  CXCL8 | 0.96 [0.55 to 1.06] | 0.73 [0.55 to 1.14]
  CXCL10 | 0.52 [0.16 to 0.79] | 0.16 [0.05 to 0.35]
  Ferritin | 0.99 [0.48 to 1.5] | 0.64 [0.39 to 1.24]
  IL-1b | 1 [0.96 to 1.86] | 1 [0.65 to 1.56]
  IL-1Ra | 1.04 [0.62 to 1.3] | 1.07 [0.59 to 1.51]
  IL-5 | 1.06 [0.86 to 1.38] | 1.09 [1 to 1.76]
  IL-6 | 0.97 [0.45 to 1.73] | 0.65 [0.19 to 1.31]

28. Other Pre Specified Outcome: Exploratory Endpoint: Change in Baseline Antiviral Immunoglobulins (IgG, IgM, IgA) at EOS
Description: Immunoglobulins measured in mg/dL
Time Frame: 28 days
Population: Change in baseline antiviral immunoglobulins were not analyzed in this study.
Arm/Group | Placebo | LSALT
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Placebo | LSALT
All-Cause Mortality (participants affected / at risk) | 0/31 | 1/30
Serious Adverse Events (participants affected / at risk) | 8/31 | 10/30
Other Adverse Events (participants affected / at risk) | 22/31 | 14/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=31) | LSALT (N=30)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus arrest (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Bacterial sepsis (Infections and infestations) | 2 | 0
Embolism (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 1
Cytokine release syndrome (Immune system disorders) | 1 | 0
Blood glucose increase (Investigations) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alkalosis (Metabolism and nutrition disorders) | 0 | 0
Hypertension (Vascular disorders) | 0 | 1
Atrial tachycardia (Cardiac disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Superinfection (Infections and infestations) | 0 | 1
Alanine aminotransferase increase (Investigations) | 0 | 1
Aspartate aminotransferase increase (Investigations) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=31) | LSALT (N=30)
Alanine aminotransferase increase (Investigations) | 9 | 5
Aspartate aminotransferase increase (Investigations) | 3 | 2
Gamma-glutamyltransferase increase (Investigations) | 2 | 0
Constipation (Gastrointestinal disorders) | 3 | 2
Toothache (Gastrointestinal disorders) | 2 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Bradycardia (Cardiac disorders) | 2 | 0
Pyrexia (General disorders) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1
Anxiety (Psychiatric disorders) | 2 | 0
Confusional state (Psychiatric disorders) | 2 | 0
Hypertension (Vascular disorders) | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-17): https://cdn.clinicaltrials.gov/large-docs/57/NCT04402957/Prot_SAP_000.pdf